CLINICAL TRIAL: NCT04989855
Title: Fruquintinib Combined With PD-1 Antibody in pMMR / MSS Locally Advanced Rectal Cancer (LARC) With High Immune Score: an Open-label, Multi-center, Phase II Clinical Trial
Brief Title: Fruquintinib Plus PD-1 Antibody in pMMR / MSS Locally Advanced Rectal Cancer (LARC) With High Immune Score
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-FLAG-C105
Record Dates: First submitted 2021-08-03; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — HMPL-013; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib plus Tislelizumab (Experimental): Fruquintinib 5mg QD d1-d14, Q3W; Tislelizumab 200mg IV Q3W d1
  Interventions: Drug: Fruquintinib plus Tislelizumab

INTERVENTIONS:
Drug: Fruquintinib plus Tislelizumab — 2 cycles of Fruquintinib(F) 5mg QD d1-d14 + Tislelizumab(T) 200mg IV d1, Q3W as preoperative therapy, and F +T after TME as postoperative therapy for 6 months

SUMMARY:
This is a prospective, one arm phase II study aimed to observe the efficacy and safety of tislelizumab combined with fruquintinib in treatment of patients with pMMR / MSS locally advanced rectal cancer with high immune score.

DETAILED DESCRIPTION:
48 patients of pMMR / MSS locally advanced rectal cancer with high immune score will be administered with tislelizumab (200mg IV d1, Q3W ) combined with fruquintinib (5mg QD d1-d14, Q3W) with a total of 2 cycles as neoadjuvant therapy. After TME, tislelizumab and fruquintinib will be given again for up to 6 months as adjuvant therapy. If the patient after neoadjuvant therapy is evaluated as SD/PD, the neoadjuvant therapy will be converted to neoadjuvant chemo-radiotherapy/chemotherapy or palliative therapy, and then the patient will be treated according to the norms of adjuvant therapy for rectal cancer if TME is performed. If the patient choose Watch & Wait when evaluated as CR, tislelizumab plus fruquintinib for at least one year is requested.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 yrs old;
2. pMMR/MSS rectal adenocarcinoma;
3. Pelvic MRI / endoscopic ultrasonography or transrectal ultrasound were used for reoperative staging: T3-4N+ with resectable tumor;
4. High immune score (Immunoscore®️ ≥3);
5. No sign of bowel obstruction, or bowel obstruction has been relieved by ostomy;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. No previous chemotherapy, radiotherapy or immunotherapy;
8. Distant metastasis was excluded by CT of chest, abdomen and pelvis before operation;
9. Able to swallow tablets;
10. Life expectancy of at least 2 years;
11. Adequate organ function;
12. Female participants of childbearing potential must be willing to use adequate contraception for the course of the study starting with the first dose of study medication through 120 days after the last PD-1 antibody dose; Male participants must agree to use adequate contraception for the course of the study starting with the first dose of study medication through 120 days after the last PD-1 antibody dose.

Exclusion Criteria:

1. Any active autoimmune disease or history of autoimmune disease;
2. Immunosuppressants, systemic or absorbable local hormones are being used to achieve the purpose of immunosuppression (dose > 10mg / day, prednisone or other effective hormones) and continue to be used within 2 weeks before enrollment;
3. History of severe allergic reaction to monoclonal antibody;
4. Subjects with untreated active brain metastasis or meningeal metastasis with clinical symptoms;
5. Suffering from hypertension and can not be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg);
6. Have previously received other PD-1 antibody therapy or other immunotherapy against PD-1 / PD-L1, or have previously received anti angiogenesis drugs;
7. There are cardiac clinical symptoms or diseases that are not well controlled, such as: (1) heart failure above NYHA grade 2 (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
8. Known hereditary or acquired bleeding and thrombotic tendency (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.) or undergoing thrombolytic or anticoagulant therapy;
9. Urine routine examination indicates that urinary protein is ≥ + +, or confirmed 24-hour urinary protein is ≥ 1.0g;
10. Significant clinical bleeding symptoms or definite bleeding tendency occurred within 3 months before enrollment, such as gastrointestinal bleeding, active bleeding, baseline fecal occult blood + + or above, or vasculitis;
11. Arteriovenous thrombosis events occurred within 6 months before enrollment, such as cerebrovascular accidents (including transient ischemic attack, intracerebral hemorrhage and cerebral infarction), deep venous thrombosis and pulmonary embolism;
12. Subjects with active infection;
13. Congenital or acquired immune deficiency (such as HIV infection) or active hepatitis (hepatitis B: HBsAg positive and HBV DNA > 104 copy number /ml; Hepatitis C: HCV antibody positive);
14. Those who participated in clinical trials of other drugs within 3 months before enrollment;
15. There was evidence of distant metastasis before operation;
16. History of pelvic or abdominal radiotherapy;
17. Any other malignant disease within the preceding 5 years with the exception of cured skin basal cell carcinoma, cervical carcinoma in situ and ovarian cancer;
18. Live vaccines were administered less than 4 weeks before the study or possibly during the study period;
19. Known or suspected allergy to the study drug or to any drug given in connection with this test;
20. In the judgment of the researcher, the subject has other circumstances that may affect the results of the study or cause the study to be forced to stop halfway.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 3 years
  Objective Response Rate

SECONDARY OUTCOMES:
3-year RFS | up to 3 years
  3-year relapse-free survival
3-year OS | up to 3 years
  3-year overall survival
Safety and Tolerability | up to 3 years
  treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- 651 Dongfeng Road East, Guangzhou, Guangdong, China